CLINICAL TRIAL: NCT01886872
Title: A Randomized Phase III Study of Bendamustine Plus Rituximab Versus Ibrutinib Plus Rituximab Versus Ibrutinib Alone in Untreated Older Patients (≥ 65 Years of Age) With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Rituximab and Bendamustine Hydrochloride, Rituximab and Ibrutinib, or Ibrutinib Alone in Treating Older Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01220; NCI-2013-01220 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ALLIANCE A041202; A041202 (Other: Alliance for Clinical Trials in Oncology); A041202 (Other: CTEP); K23CA178183 (NIH); R01CA183444 (NIH); U10CA031946 (NIH); U10CA180821 (NIH)
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Results first posted 2019-12-30 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-06

CONDITIONS: Stage I Chronic Lymphocytic Leukemia; Stage II Chronic Lymphocytic Leukemia; Stage III Chronic Lymphocytic Leukemia; Stage IV Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; Specimen Handling; Biopsy; ibrutinib; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (rituximab, bendamustine hydrochloride) (Active Comparator): Patients receive rituximab IV on day 1 (day 0 course 1) and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover to Arm II. Additionally, patients undergo bone marrow aspiration and biopsy, blood sample collection, and CT throughout the study.
  Interventions: Drug: Bendamustine Hydrochloride; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Biological: Rituximab
- Arm II (ibrutinib) (Experimental): Patients receive ibrutinib PO daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow aspiration and biopsy, blood sample collection, and CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm III (ibrutinib, rituximab) (Experimental): Patients receive ibrutinib as in Arm II. Patients receive rituximab IV on days 1, 8, 15, and 22 of course 2 and on day 1 of courses 3-6. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Additionally, patients undergo bone marrow aspiration and biopsy, blood sample collection, and CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Procedure: Computed Tomography; Drug: Ibrutinib; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Biological: Rituximab

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — Given IV
  Other Names: Belrapzo; Bendamustin Hydrochloride; Bendeka; CEP 18083; CEP-18083; CEP18083; Cytostasan Hydrochloride; Levact; Ribomustin; SyB L-0501; Treakisym; Treanda; VIVIMUSTA
  Arms: Arm I (rituximab, bendamustine hydrochloride)
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA 032765; CRA-032765; CRA032765; Imbruvica; PCI 32765; PCI-32765; PCI32765
  Arms: Arm II (ibrutinib); Arm III (ibrutinib, rituximab)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
  Arms: Arm I (rituximab, bendamustine hydrochloride); Arm III (ibrutinib, rituximab)

SUMMARY:
This randomized phase III trial studies rituximab with bendamustine hydrochloride or ibrutinib to see how well they work compared to ibrutinib alone in treating older patients with previously untreated chronic lymphocytic leukemia. Rituximab is a monoclonal antibody that may interfere with the ability of cancer cells to grow and spread. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Chemotherapy drugs, such as bendamustine hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. It is not yet known whether rituximab with bendamustine hydrochloride may work better than rituximab and ibrutinib or ibrutinib alone in treating chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine whether progression free survival (PFS) is superior after therapy with bendamustine hydrochloride (bendamustine) in combination with rituximab, ibrutinib alone, or ibrutinib in combination with rituximab in patients age 65 or older with previously untreated chronic lymphocytic leukemia (CLL).

SECONDARY OBJECTIVES:

I. To determine 2-year PFS in each of the three treatment arms. II. To determine which treatment arm produces superior overall survival (OS). III. To determine the complete response (CR) rate, complete and nodular partial response (CR/nPR) rate, and overall response (PR+nPR+CR) rate (ORR) among the three treatment arms and compare these arms.

IV. To determine the impact of minimal residual disease (MRD)-negative disease at time of CR documentation and at 2 years on PFS and OS in each of the treatment arms.

V. To determine duration of response after each of the three treatments and compare these treatment arms.

VI. To determine toxicity and tolerability of the three treatment regimens. VII. To determine response and PFS of patients initially on the bendamustine in combination with rituximab arm who cross over to ibrutinib.

OTHER PRE-SPECIFIED OBJECTIVES:

I. To determine whether baseline cytogenetic markers, Zap-70 methylation, IgVH mutational status, or select deoxyribonucleic acid (DNA) mutations predict outcomes or time to response in these three arms.

II. To determine whether local fluorescence in situ hybridization (FISH) results for del(11q22.3) and del(17p13.1) are consistent with central analysis.

III. To determine whether baseline micro ribonucleic acid (RNA) and gene expression markers are correlated with clinical outcomes of interest (e.g. progression-free and alive at 2 years versus not), as well as to explore changes in microRNA expression from baseline to post-treatment time points, with a focus on those with persistent lymphocytosis and relapse.

IV. To determine whether eradication of MRD predicts longer duration of response with standard therapy and ibrutinib-based regimens.

V. To describe the baseline functional status, comorbid medical conditions, and number of medications of older CLL patients who meet criteria for therapy.

VI. To determine how functional status changes with therapy using baseline to 3-month evaluation and end-of-study/2-year evaluation; to determine whether this change is different among the treatment groups.

VII. To determine whether geriatric assessment variables known to be associated with chemotherapy toxicity in other disease groups can also predict therapy-associated toxicity in the CLL population.

VIII. To assess whether the FCGR3A polymorphism (rs396991) is correlated with depth of response (MRD status) to ibrutinib plus rituximab after 6 cycles, with secondary endpoints CR rate, rapidity of response, and progression-free survival (PFS).

IX. To assess whether C1QA polymorphism (rs172378) is correlated with MRD status, CR rate, rapidity of response, and PFS.

OUTLINE: Patients are randomized to 1 of 3 treatment arms.

ARM I: Patients receive rituximab intravenously (IV) on day 1 (day 0 course 1) and bendamustine hydrochloride IV over 30 minutes on days 1-2. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover to Arm II.

ARM II: Patients receive ibrutinib orally (PO) daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM III: Patients receive ibrutinib as in Arm II. Patients receive rituximab IV on days 1, 8, 15, and 22 of course 2 and on day 1 of courses 3-6. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Additionally, patients undergo bone marrow aspiration and biopsy, blood sample collection, and computed tomography (CT) throughout the study.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* PRE-REGISTRATION (STEP 0)
* All patients are REQUIRED to be pre-registered to A041202 in order to submit peripheral blood to the Alliance Hematologic Malignancy Biorepository (HEME) for central Zap-70 methylation. This specimen submission is mandatory prior to registration as results will be used for stratification
* REGISTRATION (STEP 1)
* Patients must be diagnosed with CLL in accordance with International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria that includes all of the following:

  * >= 5 x 10^9 B lymphocytes (5000/uL) in the peripheral blood
  * On morphologic review, the leukemic cells must be small mature lymphocytes, and prolymphocytes must not exceed 55% of the blood lymphocytes
  * CLL cells on immunophenotype (performed locally) must reveal a clonal B-cell population, which express the B cell surface markers of CD19 and CD20, as well as the T-cell antigen CD5; patients with bright surface immunoglobulin expression or lack of CD23 expression in > 10% of cells must lack t(11;14) translocation by interphase cytogenetics
* Patients must be intermediate or high-risk Rai stage CLL

  * Intermediate risk (formerly Rai stage I/II) is defined by lymphocytosis plus enlarged lymph nodes at any site, with or without hepatomegaly or splenomegaly
  * High risk (formerly Rai stage III/IV) is defined by lymphocytosis with or without enlarged nodes and spleen plus disease-related anemia (hemoglobin < 11 g/dL) or thrombocytopenia (platelet count < 100 x 10^9/L) that is not attributable to autoimmune hemolytic anemia or thrombocytopenia
* Patients must meet criteria for treatment as defined by IWCLL 2008 guidelines which includes at least one of the following criteria:

  * Evidence of marrow failure as manifested by the development or worsening of anemia or thrombocytopenia (not attributable to autoimmune hemolytic anemia or thrombocytopenia)
  * Massive (>= 6 cm below the costal margin), progressive or symptomatic splenomegaly
  * Massive nodes (>= 10 cm) or progressive or symptomatic lymphadenopathy
  * Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy
  * Constitutional symptoms, which include any of the following:

    * Unintentional weight loss of 10% or more within 6 months
    * Significant fatigue
    * Fevers > 100.5 degrees F for 2 weeks or more without evidence of infection
    * Night sweats > 1 month without evidence of infection
* Prior treatment

  * Patients must not have had prior therapy for CLL (except palliative steroids or treatment of autoimmune complications of CLL with rituximab or steroids)
  * Treatment with rituximab and/or high dose corticosteroids for autoimmune complications of CLL must be complete at least 4 weeks prior to enrollment; palliative steroids must be at a dose not higher than 20 mg/day of prednisone or equivalent corticosteroid at the time of registration
* Age >= 65 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients with active hepatitis B defined by hepatitis B surface antigen positivity or core antibody positivity in the presence of hepatitis B DNA are not eligible for this study; patients with a positive hepatitis B core antibody but with negative hepatitis B DNA may participate, but must have hepatitis serologies and hepatitis B DNA monitored periodically by the treating physician

  * Intravenous immunoglobulin (IVIG) can cause a false positive hepatitis B serology; if patients receiving routine IVIG have core antibody or surface antigen positivity without evidence of active viremia (negative hepatitis B DNA) they may still participate in the study, but should have hepatitis serologies and hepatitis B DNA monitored periodically by the treating physician
* Patients must not be receiving active systemic anticoagulation with heparin or warfarin; patients must be off warfarin therapy for at least 30 days prior to enrollment
* Patients with class III or class IV heart failure by New York Heart Association, those with unstable angina, and those with uncontrolled arrhythmia are not eligible
* Patients who have had a myocardial infarction, intracranial bleed, or stroke within the past 6 months are not eligible
* Patients with known human immunodeficiency virus (HIV) are eligible if their CD4 count is >= 350 cells/mm^3 and if they are not taking prohibited CYP-interacting medications
* Patients must not have any history of Richter's transformation or prolymphocytic leukemia (prolymphocytes in blood > 55%)
* Patients must not require more than 20 mg prednisone or equivalent corticosteroid daily
* Patients must not have uncontrolled active systemic infection requiring intravenous antibiotics
* Patients must not have continued requirement for therapy with a strong cytochrome P450 3A4/5 (CYP3A4/5) inhibitor or inducer
* Patients must not have a known allergy to mannitol
* Patients must not have prior significant hypersensitivity to rituximab (not including infusion reactions)
* Patients may not have had major surgery within 10 days of enrollment, or minor surgery within 7 days of enrollment; examples of minor surgery include dental surgery, insertion of a venous access device, skin biopsy, or aspiration of a joint; the decision about whether a surgery is major or minor can be made at the discretion of the treating physician
* Absolute neutrophil count (ANC) >= 1,000/uL unless due to bone marrow involvement
* Aspartate aminotransferase (AST) or alanine aminotransferase (AST) =< 2.5 x upper limits of normal except if due to disease infiltration of the liver
* Bilirubin =< 1.5 x upper limits of normal (unless due to liver involvement, hemolysis, or Gilbert's disease)
* Creatinine clearance >= 40 mL/min

  * To be calculated by modified Cockcroft-Gault formula
* Platelet count (untransfused) >= 30,000/uL

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 547 (Actual)
Dates: Start 2014-01-15 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2026-06-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Woyach, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (940):
- United States (920):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Regional Hospital, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Onvida Health Yuma Medical Center, Yuma, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - John Muir Medical Center-Concord, Concord, California
  - Sutter Davis Hospital, Davis, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente-Fresno, Fresno, California
  - Marin Cancer Care Inc, Greenbrae, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente South Bay, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente West Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente Sacramento Medical Center, Sacramento, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Saint Helena Hospital, St. Helena, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Northbay Cancer Center, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Presbyterian Intercommunity Hospital, Whittier, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Kaiser Permanente-Franklin, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Saint Joseph Hospital - Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western States Cancer Research NCORP, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - National Jewish Health-Western Hematology Oncology, Golden, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Greenwood Village, Greenwood Village, Colorado
  - Kaiser Permanente-Rock Creek, Lafayette, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Kaiser Permanente-Lone Tree, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Intermountain Health Lutheran Hospital, Wheat Ridge, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Veterans Affairs Connecticut Healthcare System-West Haven Campus, West Haven, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - AdventHealth Altamonte, Altamonte Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - AdventHealth Kissimmee, Kissimmee, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - AdventHealth Medical Group Urology at Orlando, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - AdventHealth East Orlando, Orlando, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Cleveland Clinic-Weston, Weston, Florida
  - AdventHealth Winter Park, Winter Park, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - John B Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Queen's Cancer Center - Pearlridge, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - OSF Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Heartland Cancer Research NCORP, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Ascension Alexian Brothers - Elk Grove Village, Elk Grove Village, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Hematology Oncology Associates of Illinois-Highland Park, Highland Park, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Duly Health and Care Joliet, Joliet, Illinois
  - Presence Saint Mary's Hospital, Kankakee, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - AMG Libertyville - Oncology, Libertyville, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - SSM Health Good Samaritan, Mount Vernon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Quincy Medical Group-Clinic, Quincy, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - North Shore Medical Center, Skokie, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Michiana Hematology Oncology PC-Crown Point, Crown Point, Indiana
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Memorial Regional Cancer Center Day Road, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Reid Health, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Physicians' Clinic of Iowa PC, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Iowa City VA Healthcare System, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Abben Cancer Center, Spencer, Iowa
  - MercyOne Waterloo Cancer Center, Waterloo, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Newman Regional Health, Emporia, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - HaysMed, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Mercy Hospital Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cotton O'Neil Cancer Center / Stormont Vail Health, Topeka, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Ochsner Health Center-Summa, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Covington, Covington, Louisiana
  - Mary Bird Perkins Cancer Center - Houma, Houma, Louisiana
  - Ochsner Medical Center Kenner, Kenner, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - York Hospital, York Village, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Saint Agnes Hospital, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - UPMC Western Maryland, Cumberland, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Northwest Hospital Center, Randallstown, Maryland
  - TidalHealth Peninsula Regional, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Beth Israel Deaconess Medical Center/Winchester Center for Cancer Care, Winchester, Massachusetts
  - UMass Memorial Medical Center - University Campus, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Huron Valley-Sinai Hospital, Commerce, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - OSF Saint Francis Hospital and Medical Group, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital-Grosse Pointe, Grosse Pointe, Michigan
  - Allegiance Health, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - McLaren Cancer Institute-Central Michigan, Mount Pleasant, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Michigan Cancer Specialists, Roseville, Michigan
  - Oakland Colon Rectal Associates, Royal Oak, Michigan
  - Cancer Care Associates PC, Royal Oak, Michigan
  - Comprehensive Medical Center PLLC, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Hematology Oncology Consultants PC-Royal Oak, Royal Oak, Michigan
  - Oakland Medical Group, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Premier Hematology Oncology Care, Sterling Heights, Michigan
  - Mitchell Folbe MD PC, Sterling Heights, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Michigan Institute of Urology-Town Center, Troy, Michigan
  - Claudia BR Herke MD PC, Troy, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Hematology Oncology Consultants PC-Troy, Troy, Michigan
  - Henry Ford Health Warren Hospital, Warren, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Luke's Hospital of Duluth, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Lake Region Healthcare Corporation-Cancer Care, Fergus Falls, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis VA Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Cloud Hospital, Saint Cloud, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Mercy Cancer Center - Cape Girardeau, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - University Health Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Mercy Infusion Center - Chippewa, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Nevada Cancer Research Foundation NCORP, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - New Hampshire Oncology Hematology PA-Concord, Concord, New Hampshire
  - Parkland Medical Center, Derry, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - LRGHealthcare-Lakes Region General Hospital, Laconia, New Hampshire
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Dartmouth Cancer Center - Manchester, Manchester, New Hampshire
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - Dartmouth Cancer Center - Nashua, Nashua, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Veterans Adminstration New Jersey Health Care System, East Orange, New Jersey
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Penn Medicine Princeton Health, Plainsboro, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Valley Health System-Hematology/Oncology, Westwood, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Hematology Oncology Associates of Central New York-Auburn, Auburn, New York
  - Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of CNY at Camillus, Camillus, New York
  - Hematology Oncology Associates of Central New York-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Garnet Health Medical Center, Middletown, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - University of Rochester, Rochester, New York
  - Hematology Oncology Associates of Central New York-Rome, Rome, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Mission Hospital, Asheville, North Carolina
  - Mountain Radiation Oncology PA, Asheville, North Carolina
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - Messino Cancer Centers, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - Transylvania Regional Hospital, Brevard, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Angel Medical Center, Franklin, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - ECU Health Oncology Kinston, Kinston, North Carolina
  - Mission Hospital McDowell, Marion, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Blue Ridge Regional Hospital, Spruce Pine, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeast Clinical Oncology Research Consortium NCORP, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Cleveland Clinic Akron General, Akron, Ohio
  - Cleveland Clinic Cancer Center Beachwood, Beachwood, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Mercy Cancer Center-Elyria, Elyria, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Landerbrook Health Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Warren Clinic Oncology-Tulsa, Tulsa, Oklahoma
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - WellSpan Medical Oncology and Hematology, Hanover, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC Jefferson Regional Radiation Oncology, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - Associates In Hematology Oncology PC-Upland, Upland, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - Miriam Hospital, Providence, Rhode Island
  - AnMed Health Cancer Center, Anderson, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - Charleston Oncology - Roper, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-North Charleston, Charleston, South Carolina
  - Bon Secours Saint Francis Hospital, Charleston, South Carolina
  - Charleston Oncology - Saint Francis, Charleston, South Carolina
  - Lowcountry Hematology Oncology PA-West Ashley, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Greenville Health System Cancer Institute-Andrews, Greenville, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Carolina Blood and Cancer Care Associates PA-Lancaster, Lancaster, South Carolina
  - Lowcountry Hematology Oncology PA-Mount Pleasant, Mt. Pleasant, South Carolina
  - Carolina Blood and Cancer Care Associates PA, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Bristol, Bristol, Tennessee
  - Erlanger Medical Center, Chattanooga, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Ballad Health Cancer Care - Kingsport, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cancer Therapy and Research Center at The UT Health Science Center at San Antonio, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - White River Junction Veteran Administration Medical Center, White River Junction, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Hematology Oncology Associates of Fredericksburg Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Centra Alan B Pearson Regional Cancer Center, Lynchburg, Virginia
  - Ballad Health Cancer Care - Norton, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Shenandoah Oncology PC, Winchester, Virginia
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - Cancer Care Center at Island Hospital, Anacortes, Washington
  - Swedish Cancer Institute-Eastside Oncology Hematology, Bellevue, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Kaiser Permanente Washington, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Downtown, Spokane, Washington
  - Evergreen Hematology and Oncology PS, Spokane, Washington
  - MultiCare Deaconess Cancer and Blood Specialty Center - Valley, Spokane Valley, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center, Huntington, West Virginia
  - Saint Mary's Medical Center, Huntington, West Virginia
  - WVUH-Berkely Medical Center, Martinsburg, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (20):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - The Moncton Hospital, Moncton, New Brunswick
  - QEII Health Sciences Centre/Nova Scotia Health Authority, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Stronach Regional Health Centre at Southlake, Newmarket, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Michael Garron Hospital, Toronto, Ontario
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - McGill University Department of Oncology, Montreal, Quebec
  - CHUM - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Derived] Woyach JA, Perez Burbano G, Ruppert AS, Miller C, Heerema NA, Zhao W, Wall A, Ding W, Bartlett NL, Brander DM, Barr PM, Rogers KA, Parikh SA, Stephens DM, Brown JR, Lozanski G, Blachly J, Nattam S, Larson RA, Erba H, Litzow M, Luger S, Owen C, Kuzma C, Abramson JS, Little RF, Dinner S, Stone RM, Uy G, Stock W, Mandrekar SJ, Byrd JC. Follow-up from the A041202 study shows continued efficacy of ibrutinib regimens for older adults with CLL. Blood. 2024 Apr 18;143(16):1616-1627. doi: 10.1182/blood.2023021959. PMID 38215395
- [Derived] Ruppert AS, Booth AM, Ding W, Bartlett NL, Brander DM, Coutre S, Brown JR, Nattam S, Larson RA, Erba H, Litzow M, Owen C, Kuzma CS, Abramson JS, Little RF, Smith SE, Stone RM, Byrd JC, Mandrekar SJ, Woyach JA. Adverse event burden in older patients with CLL receiving bendamustine plus rituximab or ibrutinib regimens: Alliance A041202. Leukemia. 2021 Oct;35(10):2854-2861. doi: 10.1038/s41375-021-01342-x. Epub 2021 Jul 17. PMID 34274940
- [Derived] Woyach JA, Ruppert AS, Heerema NA, Zhao W, Booth AM, Ding W, Bartlett NL, Brander DM, Barr PM, Rogers KA, Parikh SA, Coutre S, Hurria A, Brown JR, Lozanski G, Blachly JS, Ozer HG, Major-Elechi B, Fruth B, Nattam S, Larson RA, Erba H, Litzow M, Owen C, Kuzma C, Abramson JS, Little RF, Smith SE, Stone RM, Mandrekar SJ, Byrd JC. Ibrutinib Regimens versus Chemoimmunotherapy in Older Patients with Untreated CLL. N Engl J Med. 2018 Dec 27;379(26):2517-2528. doi: 10.1056/NEJMoa1812836. Epub 2018 Dec 1. PMID 30501481
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive. — https://nctn-data-archive.nci.nih.gov/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 644 patients screened, 52 did not meet eligibility criteria, 19 did not register per Investigator decision, 16 did not register per patient decision, and 10 did not register for other reasons; these patients are thus excluded from the study before randomization.
Groups:
- Arm A (Rituximab, Bendamustine Hydrochloride): Patients receive rituximab 375 mg/m2 IV on day 0 of course 1 and ritixumab 500 mg/m2 IV on day 1 of courses 2-6. Patients receive bendamustine hydrochloride 90 mg/m2 IV over 30 minutes on days 1-2 of courses 1-6. Courses repeat every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients experiencing disease progression may crossover to Arm B.
- Arm B (Ibrutinib): Patients receive ibrutinib 420mg PO daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm C (Ibrutinib, Rituximab): Patients receive ibrutinib as in Arm B. Patients receive rituximab 375 mg/m2 IV on days 1, 8, 15, and 22 of course 2 and on day 1 of courses 3-6. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Started (Registered/Randomized) | 183 | 182 | 182
Evaluable for Secondary Endpoints | 183 | 182 | 182
Evaluable for Adverse Events (All Patients who Started Therapy) | 176 | 180 | 181
Crossover Cohort (Arm A to Arm B) | 30 | 0 | 0
Completed (All Eligible Patients Evaluable for the Primary Endpoint) | 176 | 178 | 170
Not Completed | 7 | 4 | 12
Not completed — Ineligible | 7 | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab) | Total
Number analyzed (Participants) | 183 | 182 | 182 | 547
Age, Continuous [Median (Full Range); unit: years] | 70 [65 to 86] | 71 [65 to 89] | 71 [65 to 86] | 71 [65 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 59 | 57 | 180
  Male | 119 | 123 | 125 | 367
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 2
  Asian | 4 | 2 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 9 | 7 | 7 | 23
  White | 167 | 169 | 173 | 509
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 1 | 7
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 98 | 87 | 86 | 271
    1 | 75 | 90 | 94 | 259
    2 | 10 | 5 | 2 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate the progression free survival distributions for each arm, with median estimates provided. Progression is defined as any one of the following: an increase in number of blood lymphocytes by >= 50% with >= 5000 B lymphocytes/mL in patients on Arm A or those on Arms 2 or 3 no longer receiving ibrutinib, >= 50% increase in the products of at least 2 lymph nodes on 2 consecutive determination 2 weeks apart, >= 50% increase in the size of the liver/spleen, transformation to a more aggressive histology, progression of any cytopenia (i.e. decrease of Hb levels > 2g/dL). Progression free survival time will be the time to either progression or death whichever occurs first.
Time Frame: Time from study entry to the time of documented disease progression or death. The analysis was event driven, performed at 2.5 years after the last patient enrolled;up to 4 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 176 | 178 | 170
months | 43 [38 to NA] — 95% Confidence interval (CI) upper limit has not been reached. | NA [NA to NA] — Median and 95% CI has not been reached. | NA [NA to NA] — Median and 95% CI has not been reached.
Statistical Analysis 1: Comparison: Arm A (Rituximab, Bendamustine Hydrochloride) vs Arm B (Ibrutinib); Arm B (Ibrutinib) versus Arm A (Rituximab, Bendamustine Hydrochloride); Test type: Superiority; p < 0.001, Log Rank — (1-sided); Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.26 to 0.58]
Statistical Analysis 2: Comparison: Arm A (Rituximab, Bendamustine Hydrochloride) vs Arm C (Ibrutinib, Rituximab); Arm C (Ibrutinib, Rituximab) versus Arm A (Rituximab, Bendamustine Hydrochloride); Test type: Superiority; p < 0.001, Log Rank — (1-sided); Hazard Ratio (HR) = 0.38, 95% CI 2-sided [0.25 to 0.59]
Statistical Analysis 3: Comparison: Arm B (Ibrutinib) vs Arm C (Ibrutinib, Rituximab); Arm C (Ibrutinib, Rituximab) versus Arm B (Ibrutinib); Test type: Superiority; p = 0.49, Log Rank — (1-sided); Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.62 to 1.62]

2. Secondary Outcome: Progression Free Survival (PFS) Rate at 2 Years
Description: The Kaplan-Meier method will be used to estimate the rate of progression free survival at 2 years in each treatment arm. Progression is defined as any one of the following: an increase in number of blood lymphocytes by >= 50%, >= 50% increase in the products of at least 2 lymph nodes on 2 consecutive determination 2 weeks apart, >= 50% increase in the size of the liver/spleen, transformation to a more aggressive histology, progression of any cytopenia (i.e. decrease of Hb levels > 2g/dL). Progression free survival time will be the time to either progression or death whichever occurs first.
Time Frame: Time from study entry to the time of documented disease progression or death, assessed up to 2 years
Population: Patient evaluable for the primary endpoint are included in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 176 | 178 | 170
percentage of patients | 74 [66 to 80] | 87 [81 to 92] | 88 [81 to 92]

3. Secondary Outcome: Overall Survival (OS) at 2 Years
Description: The Kaplan-Meier method will be used to estimate the rate of overall survival at 2 years in each treatment arm. OS will be measured from the date of registration to the date of the event (i.e., death) or the date of last follow-up to evaluate that event. Patients who are event-free at their last follow-up evaluation will be censored at that time point.
Time Frame: From the date of registration to the date of death, assessed up to 2 years
Population: Intent-to-treat analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 183 | 182 | 182
percentage of patients | 95 [91 to 98] | 90 [85 to 94] | 94 [89 to 97]

4. Secondary Outcome: Duration of Response (DOR) (Complete Response [CR], CCR, Nodular Partial Response [nPR], Partial Response [PR], and PRL)
Description: The Kaplan-Meier method will be used to estimate median DOR. DOR is the time from first objective status to progression or death. CR requires all of the following: absence of lymphadenopathy > 1.5 cm on physical exam/CT scan, no hepatomegaly/splenomegaly on physical exam, no clonal B-cells in the blood, Normal CBC, bone marrow aspirate & biopsy must be normocellular for age. PR requires >= 50% decrease in peripheral lymphocyte count from pre-treatment value, >= 50% reduction in lymphadenopathy, and/or ≥ 50% reduction in splenomegaly/hepatomegaly. CR with exception of having bone marrow lymphoid CLL nodules will be considered a nodular PR (nPR). CR with exception of not having a bone marrow biopsy performed will be considered a clinical CR (CCR). PR with the exception of having less than a 50% reduction in peripheral lymphocyte count will be considered a PR except persistent lymphocytosis (PRL).
Time Frame: From the date of first response until progression or death, performed at 2.5 years after the last patient enrolled; up to 4 years.
Population: Intent-to-treat analysis population achieving objective response
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 138 | 169 | 171
months | 50 [40 to NA] — 95% Confidence interval (CI) upper limit has not been reached. | NA [NA to NA] — Median and 95% CI has not been reached. | NA [NA to NA] — Median and 95% CI has not been reached.

5. Secondary Outcome: Percentage of Patients Achieving Any Response to Treatment (Overall Response Rate [ORR] [Complete Response [CR], CCR, Nodular Partial Response [nPR], Partial Response [PR], and PRL])
Description: Complete response (CR) requires all of the following: absence of lymphadenopathy >1.5 cm on physical exam/CT scan, no hepatomegaly/splenomegaly on physical exam, no clonal B-cells in the blood, Normal CBC, bone marrow aspirate & biopsy must be normocellular for age. Partial response (PR) requires >= 50% decrease in peripheral lymphocyte count from pre-treatment value, >= 50% reduction in lymphadenopathy, and/or ≥ 50% reduction in splenomegaly/hepatomegaly. CR with exception of having bone marrow lymphoid CLL nodules will be considered a nodular PR (nPR). CR with exception of not having a bone marrow biopsy performed will be considered a clinical CR (CCR). PR with the exception of having less than a 50% reduction in peripheral lymphocyte count will be considered a PR except persistent lymphocytosis (PRL).Overall response rate and corresponding exact binomial 95% CI provided.
Time Frame: Performed at 2.5 years after the last patient enrolled;up to 4 years.
Population: Intent-to-treat analysis population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 183 | 182 | 182
percentage of patients | 75 [69 to 81] | 93 [88 to 96] | 94 [89 to 97]

6. Secondary Outcome: Percentage of Patients Achieving a Biopsy-proven Complete Response (CR)
Description: Complete response (CR) requires all of the following: absence of lymphadenopathy > 1.5 cm on physical exam/CT scan, no hepatomegaly or splenomegaly on physical exam, no clonal B-cells in the blood, Normal CBC, bone marrow aspirate and biopsy must be normocellular for age. Complete response rate and corresponding exact binomial 95% confidence intervals provided.
Time Frame: Performed at 2.5 years after the last patient enrolled; up to 4 years.
Population: Intent-to-treat analysis population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 183 | 182 | 182
percentage of patients | 26 [20 to 33] | 7 [4 to 12] | 12 [8 to 18]

7. Secondary Outcome: Percentage of Patients Achieving Complete (CR and CCR) or Nodular Partial Response (nPR)
Description: Complete response (CR) requires all of the following: absence of lymphadenopathy > 1.5 cm on physical exam/CT scan, no hepatomegaly or splenomegaly on physical exam, no clonal B-cells in the blood, Normal CBC, bone marrow aspirate and biopsy must be normocellular for age. CR with exception of having bone marrow lymphoid CLL nodules will be considered a nodular PR (nPR). CR with exception of not having a bone marrow biopsy performed will be considered a clinical CR (CCR). Response rate and corresponding exact binomial 95% confidence intervals provided.
Time Frame: Performed at 2.5 years after the last patient enrolled; up to 4 years.
Population: Intent-to-treat analysis population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 183 | 182 | 182
percentage of patients | 33 [27 to 41] | 10 [6 to 16] | 23 [17 to 30]

8. Secondary Outcome: Percentage of Patients Who Attain Minimal Residual Disease (MRD) Negative Status
Description: Estimated using the number of patients who achieve minimal residual disease divided by the total number randomized to that treatment arm. Corresponding exact binomial 95% confidence intervals for MRD rates will be calculated.
Time Frame: Cycle 9 Day 1 Evaluation
Population: Intent-to-treat analysis population
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 183 | 182 | 182
percentage of patients | 8 [5 to 13] | 1 [0.1 to 3] | 4 [2 to 8]

9. Secondary Outcome: The Rate of Grade 3, 4, or 5 Treatment-related Non-hematologic Adverse Events (Toxicities)
Description: The rate of grade 3, 4, or 5 treatment-related non-hematologic adverse events (toxicities) by arm; excludes adverse events occurring post-crossover for patients in Arm A
Time Frame: Performed at 2.5 years after the last patient enrolled; up to 4 years.
Population: Patients who started treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab)
Number analyzed (Participants) | 176 | 180 | 181
percentage of patients | 41 | 48 | 39

10. Other Pre Specified Outcome: Geriatric Functional Status (Optional)
Description: Assessed using the Older Americans' Resources and Services Multidimensional Functional Assessment Questionnaire, Activities of Daily Living, Medical Outcomes Study physical functioning, Karnofsky performance status rated by a health care professional, Karnofsky performance status rated by the patient, timed "Up and Go", and number of falls in the last six months.
Time Frame: Performed at 2.5 years after the last patient enrolled
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Performed at 2.5 years after the last patient enrolled; up to 4 years.
Description: Patients who started treatment AND submitted at least one Adverse Events Form are included below.
Groups:
- Arm B Crossover: Arm A patients experiencing disease progression crossover to Arm B.
Arm/Group | Arm A (Rituximab, Bendamustine Hydrochloride) | Arm B (Ibrutinib) | Arm C (Ibrutinib, Rituximab) | Arm B Crossover
All-Cause Mortality (participants affected / at risk) | 15/176 | 24/180 | 22/181 | 2/27
Serious Adverse Events (participants affected / at risk) | 87/176 | 112/180 | 108/181 | 16/27
Other Adverse Events (participants affected / at risk) | 176/176 | 180/180 | 181/181 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rituximab, Bendamustine Hydrochloride) (N=176) | Arm B (Ibrutinib) (N=180) | Arm C (Ibrutinib, Rituximab) (N=181) | Arm B Crossover (N=27)
Anemia (Blood and lymphatic system disorders) | 6 (6) | 9 (13) | 6 (7) | 2 (4)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (14) | 3 (4) | 1 (1) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 19 (23) | 8 (11) | 2 (4)
Atrial flutter (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (1) | 5 (6) | 3 (4) | 0 (0)
Heart failure (Cardiac disorders) | 2 (2) | 5 (6) | 5 (6) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 2 (2) | 1 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 3 (4) | 1 (1) | 1 (1)
Pericardial tamponade (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 5 (6) | 6 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Death NOS (General disorders) | 6 (6) | 8 (8) | 7 (7) | 1 (1)
Edema face (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 4 (5) | 7 (7) | 0 (0)
Fever (General disorders) | 16 (19) | 4 (4) | 7 (7) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Infusion related reaction (General disorders) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Sudden death NOS (General disorders) | 2 (2) | 5 (5) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Anaphylaxis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Encephalitis infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 3 (3) | 4 (4) | 5 (5) | 1 (1)
Joint infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 6 (6) | 8 (9) | 12 (17) | 1 (1)
Meningitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 8 (8) | 5 (5) | 8 (9) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 6 (7) | 9 (9) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 6 (8) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 4 (6) | 2 (2) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
CPK increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (13) | 0 (0) | 2 (2) | 0 (0)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 15 (17) | 10 (11) | 11 (16) | 1 (2)
Platelet count decreased (Investigations) | 5 (6) | 3 (3) | 6 (6) | 1 (1)
Weight gain (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 3 (3) | 0 (0) | 3 (3) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 5 (5) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 16 (21) | 20 (33) | 28 (39) | 7 (10)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 3 (5) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7) | 4 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 9 (10) | 3 (4) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4 (5) | 3 (3) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (7) | 4 (4) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 6 (6) | 6 (6) | 1 (1)
Hypotension (Vascular disorders) | 6 (6) | 0 (0) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Rituximab, Bendamustine Hydrochloride) (N=176) | Arm B (Ibrutinib) (N=180) | Arm C (Ibrutinib, Rituximab) (N=181) | Arm B Crossover (N=27)
Anemia (Blood and lymphatic system disorders) | 148 (511) | 134 (743) | 131 (756) | 20 (118)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 7 (15) | 7 (14) | 4 (11) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4) | 15 (43) | 12 (23) | 2 (8)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 0 (0) | 2 (7) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Aortic valve disease (Cardiac disorders) | 2 (4) | 0 (0) | 1 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 18 (41) | 18 (45) | 4 (17)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 5 (6) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 2 (2) | 2 (3) | 2 (2) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 3 (11) | 2 (2) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (5) | 1 (3) | 1 (4)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (6) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 9 (15) | 7 (14) | 0 (0)
Paroxysmal atrial tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 3 (18) | 5 (7) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 2 (10) | 1 (10) | 2 (2) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 1 (3) | 1 (15) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 4 (4) | 5 (17) | 2 (9) | 2 (2)
Cataract (Eye disorders) | 1 (1) | 2 (6) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 3 (3) | 1 (1) | 3 (4) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 4 (14) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 3 (8) | 5 (7) | 1 (1)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Glaucoma (Eye disorders) | 0 (0) | 1 (6) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (5) | 0 (0) | 0 (0)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Scleral disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 0 (0) | 0 (0) | 3 (7) | 1 (5)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 19 (36) | 4 (4) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 3 (6) | 0 (0) | 0 (0) | 0 (0)
Bloating (Gastrointestinal disorders) | 1 (1) | 2 (15) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (4) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 33 (73) | 11 (42) | 28 (51) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 57 (95) | 95 (410) | 98 (453) | 12 (58)
Dry mouth (Gastrointestinal disorders) | 5 (9) | 7 (37) | 9 (33) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 30 (71) | 55 (225) | 73 (311) | 8 (42)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (2) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (6) | 1 (4) | 2 (2) | 0 (0)
Gastric hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 2 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 8 (26) | 7 (12) | 1 (5)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 6 (21) | 9 (19) | 5 (10) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (8) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (6) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 11 (14) | 26 (79) | 17 (53) | 1 (1)
Nausea (Gastrointestinal disorders) | 62 (134) | 25 (65) | 35 (50) | 2 (3)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral hemorrhage (Gastrointestinal disorders) | 1 (3) | 2 (2) | 1 (2) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 2 (6) | 4 (6) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (6) | 1 (2) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 14 (20) | 7 (9) | 15 (19) | 0 (0)
Chills (General disorders) | 22 (27) | 2 (2) | 11 (13) | 0 (0)
Edema face (General disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 41 (76) | 89 (383) | 96 (420) | 8 (23)
Fatigue (General disorders) | 158 (578) | 150 (1165) | 158 (1210) | 25 (167)
Fever (General disorders) | 21 (24) | 5 (5) | 5 (5) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 4 (9) | 4 (5) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (7) | 11 (23) | 13 (23) | 3 (4)
Infusion related reaction (General disorders) | 73 (97) | 0 (0) | 24 (24) | 0 (0)
Injection site reaction (General disorders) | 3 (7) | 0 (0) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 3 (7) | 1 (2) | 0 (0)
Malaise (General disorders) | 4 (5) | 2 (5) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 3 (3) | 3 (3) | 6 (9) | 0 (0)
Pain (General disorders) | 4 (4) | 3 (6) | 12 (17) | 1 (5)
Cholecystitis (Hepatobiliary disorders) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 11 (12) | 5 (5) | 10 (18) | 1 (5)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 4 (7) | 0 (0) | 1 (1) | 1 (2)
Serum sickness (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Duodenal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hepatitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 7 (9) | 7 (12) | 13 (18) | 1 (1)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 8 (11) | 5 (5) | 9 (9) | 1 (2)
Lymph gland infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (4) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Papulopustular rash (Infections and infestations) | 0 (0) | 1 (1) | 1 (3) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 3 (3) | 2 (10) | 0 (0)
Penile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis infective (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 5 (12) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 7 (8) | 7 (22) | 14 (19) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 9 (9) | 8 (10) | 14 (23) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 12 (13) | 9 (13) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 24 (43) | 117 (724) | 114 (738) | 14 (68)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 7 (8) | 4 (6) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (11) | 14 (30) | 6 (13) | 0 (0)
Alkaline phosphatase increased (Investigations) | 6 (16) | 10 (27) | 9 (20) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 9 (21) | 16 (28) | 7 (12) | 0 (0)
Blood bilirubin increased (Investigations) | 9 (27) | 21 (54) | 28 (119) | 1 (4)
CD4 lymphocytes decreased (Investigations) | 2 (8) | 0 (0) | 0 (0) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 14 (24) | 18 (74) | 23 (82) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
GGT increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hemoglobin increased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other, specify (Investigations) | 6 (7) | 8 (13) | 8 (13) | 2 (4)
Lymphocyte count decreased (Investigations) | 48 (232) | 12 (30) | 24 (62) | 7 (14)
Lymphocyte count increased (Investigations) | 17 (22) | 42 (192) | 30 (80) | 10 (22)
Neutrophil count decreased (Investigations) | 128 (356) | 61 (143) | 68 (178) | 14 (41)
Platelet count decreased (Investigations) | 138 (490) | 129 (995) | 131 (956) | 19 (104)
Urine output decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight gain (Investigations) | 1 (2) | 4 (7) | 7 (23) | 0 (0)
Weight loss (Investigations) | 13 (26) | 10 (25) | 14 (30) | 0 (0)
White blood cell decreased (Investigations) | 54 (175) | 8 (12) | 17 (37) | 2 (2)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 25 (35) | 20 (49) | 23 (40) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 1 (1) | 3 (6) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (5) | 6 (9) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 13 (31) | 16 (37) | 10 (38) | 1 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 6 (9) | 12 (25) | 7 (13) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 4 (6) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 8 (23) | 4 (6) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (9) | 11 (19) | 10 (24) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 13 (17) | 9 (17) | 7 (8) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 5 (6) | 6 (14) | 8 (13) | 2 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4) | 5 (11) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 9 (10) | 7 (11) | 12 (34) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 2 (8) | 3 (4) | 1 (2)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 6 (10) | 1 (1) | 1 (1) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (7) | 22 (84) | 26 (79) | 2 (4)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (8) | 2 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (10) | 9 (16) | 10 (15) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (3) | 1 (2) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (5) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (7) | 4 (5) | 9 (22) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (5) | 2 (2) | 0 (0)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 3 (13) | 14 (51) | 14 (44) | 0 (0)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (18) | 13 (49) | 25 (64) | 4 (7)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (5) | 3 (7) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9) | 22 (37) | 16 (24) | 1 (3)
Soft tissue necrosis lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (7) | 5 (9) | 5 (11) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 1 (4) | 0 (0)
Concentration impairment (Nervous system disorders) | 0 (0) | 2 (6) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 47 (86) | 70 (236) | 72 (248) | 10 (29)
Dysesthesia (Nervous system disorders) | 1 (2) | 0 (0) | 1 (7) | 0 (0)
Dysgeusia (Nervous system disorders) | 16 (30) | 7 (22) | 6 (10) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 7 (22) | 16 (39) | 16 (27) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 4 (7) | 3 (12) | 1 (3)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) | 2 (6) | 4 (6) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 1 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 9 (24) | 12 (31) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 2 (3) | 0 (0) | 0 (0)
Radiculitis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Spasticity (Nervous system disorders) | 0 (0) | 2 (2) | 2 (13) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 3 (3) | 3 (4) | 3 (5) | 0 (0)
Transient ischemic attacks (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 7 (14) | 3 (6) | 5 (9) | 0 (0)
Confusion (Psychiatric disorders) | 4 (4) | 5 (5) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (8) | 5 (17) | 2 (5) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (4) | 15 (35) | 8 (13) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (8) | 2 (5) | 6 (21) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1) | 10 (22) | 10 (18) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 3 (5) | 4 (16) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 4 (5) | 1 (3) | 3 (3) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (4) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 2 (4) | 1 (1) | 2 (3) | 0 (0)
Urinary urgency (Renal and urinary disorders) | 1 (3) | 1 (4) | 1 (2) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (4) | 1 (8) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (9) | 2 (2) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 74 (153) | 98 (342) | 107 (492) | 16 (66)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (39) | 22 (62) | 23 (45) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (17) | 17 (47) | 1 (6)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (3) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Laryngopharyngeal dysesthesia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (7) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (5) | 3 (3) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (4) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 4 (4) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (6) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (7) | 6 (14) | 2 (7) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (7) | 8 (26) | 10 (27) | 1 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (12) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (7) | 2 (2) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (7) | 6 (9) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periorbital edema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (11) | 10 (16) | 12 (15) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (11) | 7 (28) | 2 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2) | 4 (9) | 5 (8) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 57 (112) | 74 (271) | 72 (212) | 7 (16)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 11 (17) | 23 (86) | 18 (37) | 3 (5)
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (12) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (5) | 0 (0)
Social circumstances - Other, specify (Social circumstances) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 2 (3) | 6 (12) | 1 (1)
Hot flashes (Vascular disorders) | 2 (3) | 3 (12) | 3 (7) | 1 (4)
Hypertension (Vascular disorders) | 81 (276) | 121 (1146) | 126 (1119) | 19 (133)
Hypotension (Vascular disorders) | 10 (11) | 0 (0) | 3 (4) | 0 (0)
Phlebitis (Vascular disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 2 (3) | 3 (3) | 2 (4) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT01886872/Prot_SAP_000.pdf